CLINICAL TRIAL: NCT06425861
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1, Single and Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Food Effect of THB335 in Healthy Participants
Brief Title: A First in Human Trial Evaluating THB335 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Third Harmonic Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THB335-101
Record Dates: First submitted 2024-05-15; First posted 2024-05-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- THB335 single dose (Experimental): Single dose of THB335 fasted
  Interventions: Drug: THB335 single dose
- THB335 fasted and fed (Experimental): Single dose of THB335 fasted and then fed
  Interventions: Drug: THB335 fasted/fed
- THB335 multiple dose (Experimental): 14 days of multiple ascending doses of THB335
  Interventions: Drug: THB335 multiple dose
- Single dose placebo (Placebo Comparator): Single dose of placebo capsule, fasted
  Interventions: Drug: Single dose placebo
- Fasted and fed placebo (Placebo Comparator): Single dose of placebo capsule fasted and then fed
  Interventions: Drug: Placebo fasted/fed
- Multiple dose placebo (Placebo Comparator): 14 days of multiple doses of placebo capsule
  Interventions: Drug: Multiple dose placebo

INTERVENTIONS:
Drug: THB335 single dose — Single dose as oral capsule
  Arms: THB335 single dose
Drug: Single dose placebo — Single dose as oral capsule
  Arms: Single dose placebo
Drug: THB335 fasted/fed — Single dose fasted and fed as oral capsule
  Arms: THB335 fasted and fed
Drug: Placebo fasted/fed — Single dose fasted and fed as oral capsule
  Arms: Fasted and fed placebo
Drug: THB335 multiple dose — Multiple ascending doses oral capsule
  Arms: THB335 multiple dose
Drug: Multiple dose placebo — Multiple doses oral capsule
  Arms: Multiple dose placebo

SUMMARY:
This study is a double blind, randomized, placebo-controlled, Phase 1 study in three parts: single ascending doses and food effect (Part 1), multiple ascending doses (Part 2) and Relative Bioavailability of Two Formulations (Part 3).

DETAILED DESCRIPTION:
THB335 is a highly potent and selective inhibitor of the receptor tyrosine kinase KIT that is expressed on mast cells.

The study will evaluate the safety, pharmacokinetics, pharmacodynamics, and food effect profile of THB335 administered orally in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* In good health, determined by no clinically significant findings from medical history, 12 lead electrocardiogram (ECG), vital sign measurements, and clinical laboratory evaluations
* Males or females, of any race, between 18 and 65 years of age, inclusive.
* Participants must understand the nature of the study and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any study related procedures
* Body weight of ≥ 50.0 kg for men and ≥ 45.0 kg for women and Body Mass Index (BMI) of 17.5-32.0 kg/m2 (inclusive) at Screening

Exclusion Criteria:

* Significant history or clinical manifestation of cancer or any metabolic, allergic, dermatological, hepatic, biliary, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* Vaccinated within 14 days prior to Day -1 or intention to receive vaccination during the study
* A positive urine drug screen/alcohol breath test
* The participant currently smokes, vapes, or uses nicotine-containing products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | Part 1 Day 1 through Day 9 (end of study), and Part 2 Day 1 through Day 29 (end of study)

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Part 1, and Part 2 on Day 1. Part 2 on Day 14
Time to Cmax (Tmax) | Part 1, and Part 2 on Day 1. Part 2 on Day 14
Area under the plasma concentration-time curve (AUC) | Part 1, and Part 2 on Day 1. Part 2 on Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — QPS Holdings LLC
Locations (1):
- QPS Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No